CLINICAL TRIAL: NCT04391907
Title: Clinical Efficacy of Intense Pulsed Light(IPL) Procedure in Dry Eye Patients With Meibomian Gland Dysfunction Prior to Cataract Surgery
Brief Title: Clinical Efficacy of Intense Pulsed Light(IPL) Procedure in Dry Eye Patient
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to the covid 19, patient recruiment is not going smoothly, so the study was canceled.
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, tae-young chung, Professor, Samsung Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019-07-016
Record Dates: First submitted 2020-05-15; First posted 2020-05-18 (Actual); Last update posted 2022-05-13 (Actual); Status verified 2022-05

CONDITIONS: Dry Eye Syndromes
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IPL group (Active Comparator): Subject who have intense pulsed light (IPL) laser 2 twice 1-6 weeks before cataract surgery
  Interventions: Procedure: IPL
- Non-IPL group (No Intervention): Subject who do not have intense pulsed light (IPL) laser before cataract surgery

INTERVENTIONS:
Procedure: IPL — Intense pulse light (IPL) laser is used for the treatment of dry eye originated from meibomian gland dysfunction. IPL laser will be performed to patients who are planned to cataract surgery to improve dry eye.
  Arms: IPL group

SUMMARY:
Clinical efficacy of Intense Pulsed Light(IPL) procedure in dry eye patients with meibomian gland dysfunction prior to cataract surgery.

DETAILED DESCRIPTION:
IPL procedure is a device used for symptom relief and treatment of dry eye syndrome caused by meibomian gland dysfunction in adults, and its safety and long-term effects have been confirmed. The purpose of this study is to determine whether this procedure before cataract surgery is effective in improving the symptoms of dry eye syndrome after cataract surgery.

ELIGIBILITY:
Inclusion Criteria:

1. A patient at the age of 21 cataract surgery
2. A patient has the visual potential of 20/25 or better in each eye after cataract removal
3. Dry eye patient by meibomian gland dysfunction
4. Written informed consent to surgery and participation in the study

Exclusion Criteria:

1. Eye damage, active eye infection
2. Uncontrolled health problem
3. Wear contact lens within one month
4. Allergic reactions of fluorescein sodium or ophtalmic anesthetic
5. Eye surgery and trauma in the last six months
6. Eye disease, structural abnormality
7. If there is a cause of vision loss other than cataracts
8. Under 20/25 expect vision
9. Under the age of 20 years of age
10. Pregnant woman and lactating woman
11. Medical conditions in which IPL is contraindicated

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-03-03 (Estimated); Primary Completion 2021-03-02 (Estimated); Study Completion 2021-03-02 (Estimated)

PRIMARY OUTCOMES:
TBUT | 3 months
  tear break-up time
meibomian gland function score | 3 months
  By expression of eyelid, scoring of expressibility and quality of meibum will be tested. Form of secretion predominantly secreted by the eight meibomian glands in the center of the lid was evaluated as follows. grade 0, clear meibum is easily expressed; grade 1, cloudy meibum is expressed with mild pressure; grade 2, cloudy meibum is expressed with more than moderate pressure; and grade 3, meibum cannot be expressed even with the hard pressure. Higher score means a worst outcome.

SECONDARY OUTCOMES:
OSDI | 3 months
  questionnaire to evaluate dry eye symptoms. OSDI grading (0 ~ 100) was as follows: normal (0-12 points), mild (13-22 points), moderate (23-32 points), or severe (33-100 points). Higher score means a worse outcome.
Corneal staining score | 3 months
  Punctate epithelial erosion of cornea will be evaluated with standard classification system(NEI score, National Eye Institute score). It divides the cornea into five sections and assigns a value from 0 (absent) to 3 (severe) to each section, based on the amount, size, and confluence of the PEE, for a maximum of 15 points. Higher score means a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Tae-Young Chung, PhD, Study Chair — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea